CLINICAL TRIAL: NCT06880549
Title: A Phase 1, Open-label, Multicenter, Dose-escalation Study of mRNA-4106 Administered Alone and in Combination With Immune Checkpoint Blockade in Participants With Solid Tumors
Brief Title: A Study of mRNA-4106 Administered Alone and in Combination With Immune Checkpoint Blockade in Participants With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-4106-P101; NCT06880536 (obsolete NCT alias)
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors
Keywords: Locally advanced; Metastatic; Relapsed or refractory solid tumor malignancies; Nivolumab/relatlimab; Oncology; Melanoma; Solid tumors
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Neoplasms; Melanoma | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Dose Escalation): mRNA-4106 Alone (Experimental): Participants will receive mRNA-4106 at a test dose as monotherapy.
  Interventions: Biological: mRNA-4106
- Arm 2 (Dose Confirmation): mRNA-4106 in Combination with Nivolumab/Relatlimab (Experimental): Participants will receive mRNA-4106 at an applicable dose in combination with nivolumab/relatlimab at a standard dose.
  Interventions: Biological: mRNA-4106; Biological: Nivolumab/Relatlimab

INTERVENTIONS:
Biological: mRNA-4106 — Intramuscular Injection
Biological: Nivolumab/Relatlimab — Intravenous infusion
  Arms: Arm 2 (Dose Confirmation): mRNA-4106 in Combination with Nivolumab/Relatlimab

SUMMARY:
The purpose of this study is to assess the safety and tolerability of mRNA-4106 administered alone and in combination with checkpoint inhibitor (CPI) therapy in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1, Monotherapy Arm: Histologically confirmed advanced or metastatic cancer (melanoma, non-small cell lung cancer (NSCLC), hepatocellular carcinoma (HCC), esophageal carcinoma, head and neck squamous cell carcinoma (HNSCC), urinary bladder cancer (UBC), colon/rectal adenocarcinomas, gastric, ovarian, cervical, and endometrial carcinomas) with measurable disease as determined by RECIST v1.1 and have completed or refused all standard therapies (no limit to prior lines of therapy). Participants must have a tumor lesion amenable to biopsy, or alternatively archival tumor tissue is acceptable as long as the collection date is within one year of the enrollment date.
* Arm 2, Combination with Nivolumab/Relatlimab Arm: Histologically confirmed unresectable or metastatic melanoma, with measurable disease as determined by RECIST v1.1 and have not had any prior therapy for this cancer in this setting (that is, first-line therapy). Note that prior adjuvant, neoadjuvant, or perioperative melanoma therapy (that is, anti-CTLA-4, anti-PD1/L1, BRAF/MEK inhibitors, or interferon) is permitted if disease recurrence did not occur within 3 months from the last treatment date.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
* Participant has adequate hematological and biological function.
* Participants who could become pregnant: negative pregnancy test within 24 hours before the first dose of study treatment.

Exclusion Criteria:

* Participant has active central nervous system tumors or metastases
* Participant has received treatment with prohibited medications/treatments (ie, concurrent anticancer therapy including other chemotherapy, hormonal anticancer therapy, biologic therapy, or immunotherapy) or investigational agents within 5 half-lives or 14 days prior to the first day of study treatment (Cycle 1 Day 1), whichever is shorter.
* Participant has required the use of immunosuppressive doses of systemic steroids or absorbed topical steroids (doses >10 mg prednisone daily equivalent) within 2 weeks before study treatment administration or currently requiring maintenance doses of >10 mg prednisone or equivalent per day.
* Participant has any plan to receive a live attenuated vaccine during study treatment or has received a live vaccine within 30 days before the first dose of study treatment.
* Participant has reversible toxicities from prior cancer therapy that have not recovered to Grade 1 or baseline. Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and prespecified laboratory values.
* Participant has any unstable or clinically significant concurrent medical/psychiatric illness or social situation that would limit compliance with study requirements or compromise the ability of the participant to provide written informed consent, per the discretion of the Investigator.
* Participant has concurrent enrollment in another clinical study (unless it is an observational noninterventional clinical study).

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2029-01-10 (Estimated); Study Completion 2029-01-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | For Arm 1: Days 1-21 and Arm 2: Days 1-28
Number of Participants With Treatment Emergent Adverse Events, Serious Adverse Events and Adverse Events of Special Interest | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - START Midwest, Grand Rapids, Michigan
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah